CLINICAL TRIAL: NCT05537766
Title: A Phase 2, Open-Label, Multicenter, Basket Study Evaluating the Efficacy of Brexucabtagene Autoleucel in Adults With Rare B-cell Malignancies (ZUMA-25)
Brief Title: Study of Brexucabtagene Autoleucel in Adults With Rare B-cell Malignancies
Acronym: ZUMA-25
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to terminate study.
Sponsor: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KT-US-568-0138; 2022-501259-10 (Other: European Medicines Agency); 2022-501260-18 (Other: European Medicines Agency); 2022-501261-46 (Other: European Medicines Agency); 2022-501262-21 (Other: European Medicines Agency)
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Relapsed/Refractory Waldenstrom Macroglobulinemia; Relapsed/Refractory Richter Transformation; Relapsed/Refractory Burkitt Lymphoma; Relapsed/Refractory Hairy Cell Leukemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Recurrence; Burkitt Lymphoma; Leukemia, Hairy Cell | interventions — brexucabtagene autoleucel; Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Substudy A (Relapsed/Refractory Waldenstrom Macroglobulinemia): Brexucabtagene Autoleucel (Experimental): Participants will receive fludarabine 30 mg/m^2/day and cyclophosphamide 500 mg/m^2/day lymphodepletion chemotherapy for 3 days followed by a single infusion of brexucabtagene autoleucel at target dose of 2 × 10^6 anti-CD19 chimeric antigen receptor (CAR) T cells/kg.
  This arm is no longer recruiting.
  Interventions: Biological: Brexucabtagene Autoleucel; Drug: Cyclophosphamide; Drug: Fludarabine
- Substudy B (Relapsed/Refractory Richter Transformation): Brexucabtagene Autoleucel (Experimental): Participants will receive fludarabine 30 mg/m^2/day and cyclophosphamide 500 mg/m^2/day lymphodepletion chemotherapy for 3 days followed by a single infusion of brexucabtagene autoleucel at target dose of 2×10^6 anti-CD19 CAR T cells/kg.
  This arm is no longer recruiting.
  Interventions: Biological: Brexucabtagene Autoleucel; Drug: Cyclophosphamide; Drug: Fludarabine
- Substudy C (Relapsed/Refractory Burkitt Lymphoma): Brexucabtagene Autoleucel (Experimental): Participants will receive fludarabine 30 mg/m^2/day and cyclophosphamide 500 mg/m^2/day lymphodepletion chemotherapy for 3 days followed by a single infusion of brexucabtagene autoleucel at a target dose of 2x10^6 anti-CD19 CAR T cells/kg.
  Interventions: Biological: Brexucabtagene Autoleucel; Drug: Cyclophosphamide; Drug: Fludarabine
- Substudy D (Relapsed/Refractory hairy cell leukemia): Brexucabtagene Autoleucel (Experimental): Participants will receive fludarabine 30 mg/m^2/day and cyclophosphamide 500 mg/m^2/day lymphodepletion chemotherapy for 3 days followed by a single infusion of brexucabtagene autoleucel at a target dose of 2 × 10^6 anti-CD19 CAR T cells/kg.
  This arm is no longer recruiting.
  Interventions: Biological: Brexucabtagene Autoleucel; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: Brexucabtagene Autoleucel — Administered intravenously
  Other Names: KTE-X19
Drug: Cyclophosphamide — Administered intravenously
Drug: Fludarabine — Administered intravenously

SUMMARY:
Master protocol: The goal of this master clinical study is to test how well the study drug, brexucabtagene autoleucel, works in participants with rare B-cell malignancies: relapsed/refractory Waldenstrom macroglobulinemia (r/r WM) (Substudy A - no longer recruiting), relapsed/refractory Richter transformation (r/r RT) (Substudy B), relapsed/refractory Burkitt lymphoma (r/r BL) (Substudy C and relapsed/refractory hairy cell leukemia (r/r HCL) (Substudy D - no longer recruiting).

DETAILED DESCRIPTION:
Master protocol: The primary objective of this study is to evaluate the efficacy of brexucabtagene autoleucel in two rare B-cell malignancies. This study will use a basket study design with separate, indication-specific substudies, to investigate r/r RT and r/r BL.

After completing the treatment period, all participants will be followed in the post-treatment follow-up period. Thereafter, participants will transition to a separate long-term follow-up study (KT-US-982-5968) to continue follow-up out to 15 years.

Substudies A and D have been early terminated by the sponsor.

ELIGIBILITY:
Key Inclusion Criteria:

All Substudies:

* Presence of toxicities due to prior therapy must be stable and recovered to Grade 1 or lower.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Adequate hematologic and end-organ function.
* Individuals of childbearing potential who engage in heterosexual intercourse must agree to use specified method(s) of contraception.

Substudy B:

* Confirmed diagnosis of chronic lymphocytic leukemia (CLL) based on International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2018 criteria with histologically confirmed Richter transformation (RT) to a diffuse large B-cell lymphoma (DLBCL) subtype.
* Relapsed or refractory disease after 1 line of therapy, defined as at least 1 of the following:

  * Refractory disease, defined as progressive disease or stable disease as best response to first-line therapy.
  * Relapsed disease, defined as complete remission to first-line therapy followed by biopsy-proven disease relapse.
* At least 1 measurable lesion based on the Lugano Classification. Lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy.

Substudy C:

* Histologically confirmed mature B-cell non-Hodgkin lymphoma (NHL) Burkitt lymphoma/leukemia.
* Relapsed or refractory disease after first-line chemoimmunotherapy, defined as 1 of the following:

  * Refractory disease, defined as progressive disease or stable disease as best response to first-line therapy; individuals who are intolerant to first-line therapy are excluded.
  * Relapsed disease, defined as complete remission to first-line therapy followed by biopsy-proven disease relapse.
* At least 1 measurable lesion based on the Lugano Classification. Lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy.

Key Exclusion Criteria:

All Substudies:

* Prior CAR therapy or treatment with any anti-CD19 therapy.
* HIV-positive patients, unless taking appropriate anti-HIV medications, having an undetectable viral load by quantitative polymerase chain reaction (qPCR) and a CD4 count > 200 cells/uL.
* Presence of detectable cerebrospinal fluid malignant cells or brain metastases.
* History of autoimmune disease (eg, Crohn's disease, rheumatoid arthritis, systemic lupus).

Substudy B:

* Diagnosis of RT not of DLBCL subtype (including, but not limited to, Hodgkin lymphoma (HL) and prolymphocytic leukemia).
* Prior allogeneic or autologous stem cell transplant < 3 months prior to screening and/or < 4 months prior to planned infusion of brexucabtagene autoleucel.
* Presence of active graft-versus-host disease following prior stem cell transplant.

Substudy C:

* Burkitt-like lymphoma with 11q aberration, high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangement, or high-grade B-cell lymphoma not otherwise specified.
* Prior allogeneic stem cell transplant < 3 months prior to screening and/or < 4 months prior to planned infusion of brexucabtagene autoleucel.
* Presence of active graft-versus-host disease following prior allogeneic stem cell transplant.
* Presence of CNS involvement. Individuals with a prior history of CNS involvement are eligible if they show a negative CSF and no involvement by imaging.

Substudies A and D have been early terminated by the sponsor.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Substudy A: Combined Rate of Complete Response (CR) and Very Good Partial Response (VGPR) Determined by Central Assessment per the Sixth International Workshop in Waldenstrom Macroglobulinemia (WM) | Up to 5 years
  Combined rate is defined as the proportion of participants who achieve either CR or VGPR.
Substudy B: Objective Response Rate (ORR) Determined by Central Assessment per the Lugano Classification | Up to 2 years
  ORR is defined as the proportion of participants who achieve a best response of either CR or partial response (PR).
Substudy C: ORR Determined by Central Assessment per the Lugano Classification | Up to 2 years
  ORR is defined as the proportion of participants who achieve a best response of either CR or PR.
Substudy D: ORR Determined by Central Assessment per the Response Criteria Described by Grever and Colleagues | Up to 5 years
  ORR is defined as the proportion of participants who achieve either CR or PR.

SECONDARY OUTCOMES:
All Substudies (Substudies A, B, C and D): Complete Response (CR) Rate Determined by Central Assessment | Up to 2 years for substudies B and C; Up to 5 years for substudies A and D
  CR rate is defined as proportion of participants who achieve CR.
All Substudies (Substudies A, B, C and D): Duration of Response (DOR) | Up to 2 years for substudies B and C; Up to 5 years for substudies A and D
  DOR is defined as time from first objective response to disease progression per indication specific response criteria or death from any cause.
All Substudies (Substudies A, B, C and D): Overall Survival (OS) | Up to 2 years for substudies B and C; Up to 5 years for substudies A and D
  OS is defined as the time from enrollment or brexucabtagene autoleucel infusion to death from any cause.
All Substudies (Substudies A, B, C and D): Progression Free Survival (PFS) | Up to 2 years for substudies B and C; Up to 5 years for substudies A and D
  PFS is defined as the time from enrollment or brexucabtagene autoleucel infusion to disease progression per indication specific response criteria or death from any cause.
All Substudies (Substudies A, B, C and D): Time to Next Treatment (TTNT) | Up to 2 years for substudies B and C; Up to 5 years for substudies A and D
  TTNT defined as the time from enrollment or brexucabtagene autoleucel infusion to the initiation of subsequent anticancer treatment.
All Substudies (Substudies A, B, C and D): Time to First Response | Up to 2 years for substudies B and C; Up to 5 years for substudies A and D
  Time to first response is defined as the time from enrollment or brexucabtagene autoleucel infusion to first objective response.
All Substudies (Substudies A, B, C and D): Time to Best Response | Up to 2 years for substudies B and C; Up to 5 years for substudies A and D
  Time to best response is defined as the time from enrollment or brexucabtagene autoleucel infusion to best objective response.
All Substudies (Substudies A, B, C and D): Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | First infusion date up to 2 years plus 30 days for substudies B and C; First infusion date up to 5 years plus 30 days for substudies A and D
All Substudies (Substudies A, B, C and D): Percentage of Participants Experiencing Clinically Significant Changes in Safety Laboratory Values | First infusion date up to 2 years plus 30 days for substudies B and C; First infusion date up to 5 years plus 30 days for substudies A and D
All Substudies (Substudies A, B, C and D): Percentage of Participants Experiencing Adverse Events (AEs) Defined as Dose Limiting Toxicities (DLTs) | First infusion date of brexucabtagene autoleucel up to 28 days
  Dose-limiting toxicity is defined as protocol-defined brexucabtagene autoleucel-related events with onset within the first 28 days following brexucabtagene autoleucel infusion.
All Substudies (Substudies A, B, C and D): Percentage of Participants With Positive Anti-brexucabtagene autoleucel Antibodies | First infusion date Up to 2 years for substudies B and C; First infusion date Up to 5 years for substudies A and D
All Substudies (Substudies A, B, C and D): Percentage of Participants With Replication-competent Retrovirus (RCR) in Peripheral Blood Mononuclear Cells (PBMCs) | Baseline, Month 12
All Substudies (Substudies A, B, C and D): Change From Baseline in the European Organisation for Research and Treatment of Cancer-Quality of Life Questionnaire-30 (EORTC QLQ-C30) Score | Baseline, up to 24 months
  The EORTC-QLQ-C30 is a multi-item questionnaire measuring the following content five (5) multi-item functional scales, six (6) multi-item symptom scales, one (1) global health status scale, and one (1) global health-related quality of life (HRQoL) each scale is measured from 0 to 100 after a linear transformation. Higher scores for functioning scales and for the Global Health Status or Global HRQoL scales indicate a higher level of functioning and a better HRQoL respectively, whereas higher scores in symptom scales represent a higher level of symptoms.
All Substudies (Substudies A, B, C and D): Changes From Baseline in the European Quality of Life Five Dimensions Five Levels Questionnaire (EQ-5D-5L) Score | Baseline, Up to 24 months
  The EQ-5D-5L questionnaire is a generic measure of health status that provides a simple descriptive profile and a single index value. The EQ-5D-5L comprises 2 components: a questionnaire covering 5 dimensions and a tariff of values based upon direct valuations of health states using a visual analog scale (VAS). Rating gets recorded on a vertical VAS in which the endpoints are labeled best imaginable health state is 100 (on the top) and worst imaginable health state is 0 (on the bottom). Higher scores of EQ VAS indicate better health.
Substudy A: ORR Determined by Central Assessment | Up to 5 years
  ORR is defined as the proportion of participants who achieve a best response of CR, VGPR, or PR.
Substudy A: Combined CR and VGPR Rate Determined by Investigator Assessment | Up to 5 years
  Combined rate is defined as the proportion of participants who achieve either CR or VGPR.
Substudy A: PR Rate Determined by Central Assessment | Up to 5 years
  PR rate is defined as proportion of participants who achieve PR.
Substudy A: VGPR Rate Determined by Central Assessment | Up to 5 years
  VGPR rate is defined as proportion of participants who achieve VGPR.
Substudy B: ORR Determined by Investigator Assessment per the Lugano Classification | Up to 2 years
  ORR is defined as the proportion of participants who achieve a best response of either CR or PR.
Substudy B: ORR Determined by Central Assessment per the Lugano Classification | Up to 2 years
  ORR is defined as the proportion of participants who achieve a best response of either CR or PR, in subgroups by clonal relationship to the underlying CLL. Clonality will be assessed by central assessment.
Substudy B: ORR Determined by Investigator per International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2018 Criteria | Up to 2 years
  ORR is defined as the proportion of participants who achieve a best response of either CR, complete response with incomplete marrow recovery (CRi) or PR.
Substudy C: ORR Determined by Investigator Assessment per the Lugano Classification | Up to 2 years
  ORR is defined as the proportion of participants who achieve a best response of either CR or PR.
Substudy D: ORR Determined by Investigator Assessment | Up to 5 years
  ORR is defined as the proportion of participants who achieve either CR or PR.

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (26):
- United States (12):
  - City of Hope (City of Hope National Medical Center), Duarte, California
  - Stanford Cancer Institute, Stanford, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Georgetown University Medical Centre, Washington D.C., District of Columbia
  - University of Iowa, Iowa City, Iowa
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Ohio State University Wexner Medical Center - James Cancer HospitalS, Columbus, Ohio
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Medical University of Vienna, Department of Internal Medicine I, Div. of Hematology, Vienna, Austria
- France (2):
  - Hopital de la Pitie Salpetriere, Paris
  - Centre hospitalier de Toulouse - Hematology department, Toulouse
- Germany (3):
  - Universitatsklinikum Koln, Cologne
  - Universitatsklinikum Heidelberg, Heidelberg
  - Universitatsklinikum Ulm, Ulm
- Italy (3):
  - IRCCS Azienda Ospedaliero - Universitaria di Bologna, Bologna
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedale di Perugia - Ospedale S. Maria della Misericordia, Perugia
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands
- Spain (3):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
- Istituto Oncologico Della Svizzera Italiana (IOSI), Bellinzona, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=KT-US-568-0138